CLINICAL TRIAL: NCT01968226
Title: An Exploratory, Phase II, Open Label, Single-Center, Non-Randomized Study Of [F-18] RGD-K5 Positron Emission Tomography (PET) In Participants With Carotid Artery Stenosis
Brief Title: TRACER RGD-K5 Carotid Plaque Imaging Study
Acronym: TRACER
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Investigator left instititution
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: K5 IND
Record Dates: First submitted 2013-10-17; First posted 2013-10-23 (Estimated); Results first posted 2017-08-10 (Actual); Last update posted 2017-09-12 (Actual); Status verified 2017-08

CONDITIONS: Carotid Artery Disease; Carotid Stenosis
Keywords: carotid artery disease; carotid stenosis; carotid endarterectomy; RDG-K5; PET imaging
MeSH Terms: conditions — Carotid Artery Diseases; Carotid Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PET imaging with [F-18] RDG-K5 (Experimental): This is an observational study of a group of individuals who all have carotid artery stenosis. The observation will be the measurement of [F-18]RGD-K5 uptake by the carotid artery plaque after intravenous administration of this radiolabeled tracer using PET imaging.
  Interventions: Drug: [F-18] RDG-K5

INTERVENTIONS:
Drug: [F-18] RDG-K5 — Up to fifteen (15) subjects with carotid stenosis >50% who are undergoing planned carotid endarterectomy will be imaged under PET with [F-18] RDG-K5
  Other Names: Radiolabeled tracer

SUMMARY:
The purpose of this study is to investigate the ability of the compound[F-18]RGD-K5, when used as a tracer during PET (positron emission tomography) imaging, to detect regions of unstable atherosclerotic plaque in the carotid artery of subjects being considered for carotid endarterectomy (CEA),and to confirm this ability through histological studies of samples of carotid artery plaques that will be collected during the planned carotid surgery.

DETAILED DESCRIPTION:
Patients will be chosen for the study based on presence of carotid artery stenosis ascertained by CTA and carotid artery ultrasound. Patients will receive and intravenous injection of the radiolabeled PET tracer,[F-18]RGD-K5, and will undergo PET imaging of their carotid arteries bilaterally. PET images will be analyzed to determine the standard uptake value (SUV) of [F-18]RGD-K5 uptake by the carotid artery plaque and this will be compared to the SUV of the background (blood pool in the aorta). This will be expressed as a target to background ratio (TBR). Investigators expect to find a significant uptake of [F-18]RGD-K5 by carotid artery palque and investigators therefore expect to find a TBR that is significantly >1. Investigators also expect to find that plaque from patients who show a TBR >1 will also be enriched for histologic markers for inflammation and angiogenesis.

ELIGIBILITY:
Inclusion Criteria:

* Participant is a female or male of any race/ethnicity >18 years old at the time of the investigational product administration
* Participant or participant's legally acceptable representative provides written informed consent
* Participant is capable of complying with study procedures
* Participant has known carotid artery stenosis of >50% luminal diameter based on carotid ultrasound or computed tomography angiography (CTA), as stated in official clinical report or as measured by PI if no quantitative assessment appears in the report, and who is deemed to be a surgical candidate for endarterectomy
* Participant has had a carotid ultrasound and/or computed tomography angiography (CTA) and the report is available for collection
* Participant has had or is scheduled to have a carotid CT angiogram for plaque localization within 60 days of signing ICF (or else scheduled CTA must be performed on a separate day and prior to the investigational PET procedure)
* Participant has consented to have an endarterectomy
* Participant will be scheduled for an investigational[F-18]RGD-K5 PET/CT scan within 4 weeks prior to endarterectomy
* Participant must have renal functions values as defined by laboratory results within the following ranges:

  * Serum creatinine ≤ 1.5 mg/dL
  * Estimated glomerular filtration rate (eGFR): ≥ 45mL/min

Exclusion Criteria:

* Female participant is nursing
* Female participant is pregnant
* Participant has been involved in an investigative, radioactive research procedure within the past 14 days
* Participant has any other condition or personal circumstance that, in the judgment of the investigator, might interfere with the collection of complete data or data quality
* Participant has a history or current evidence of any condition, therapy, lab abnormality that, in the opinion of the study investigator or treating physicians might confound the results of the study or poses an additional risk to the participants by their participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Balaji Tamarappoo, MD, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PET Imaging With [F-18] RDG-K5
Started | 3
Completed | 1
Not Completed | 2
Not completed — [F-18] RDG-K5 was not available | 2

BASELINE CHARACTERISTICS:
Population: Due to trial termination, no subject analysis was completed
Arm/Group | PET Imaging With [F-18] RDG-K5
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants] — No subject data analyzed Population: Study terminated, no subject data analyzed
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Target to Background Ratio (TBR)
Description: To assess uptake of [F-18]RGD-K5 by carotid plaque with PET/CT imaging (which will be expressed as a target to background ratio (TBR) of the standard uptake value (SUV)) in participants prior to carotid endarterectomy. The TBR of [F-18]RGD-K5 in the plaque will serve as a surrogate marker of plaque inflammation in participants being considered for carotid endarterectomy.
Time Frame: Baseline
Population: no subject analysis done
Arm/Group | PET Imaging With [F-18] RDG-K5
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | PET Imaging With [F-18] RDG-K5
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes